CLINICAL TRIAL: NCT05038176
Title: Improving the Diabetic Health of Black Men (MANUP-NC): MANUP-NC Feasibility Trial
Brief Title: Improving the Diabetic Health of Black Men: MANUP Feasibility Trial
Acronym: MANUP-NC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina Central University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NCCU
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2; Coping Behavior; Self Efficacy; Masculinity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Masculinity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention group (AI) (Experimental): The active intervention group (AI) receiving the active treatment (MANUP intervention) which include diabetes education, diabetes support with a focus on coping techniques (based on John Henryism concepts), physical activity engagement and motivational text messages.
  Interventions: Behavioral: MANUP
- Delayed intervention group (DI) (Active Comparator): DI participants will only receive motivational text-messages. They will then "flip" and receive full intervention after the AI group has completed the program.
  Interventions: Behavioral: MANUP

INTERVENTIONS:
Behavioral: MANUP — Intervention will include diabetes education, diabetes support with a focus on coping techniques (based on John Henryism concepts), physical activity engagement and motivational text messages.

SUMMARY:
Many Black Americans continue to be suffer from diabetes especially Black men. Although previous diabetes efforts have reduced overall disease burden, they have failed to eliminate racial and geographic disparities. The story of John Henry, the "steel-drivin' man" represents strength and self-determination among Black Men. But often these traits lead men to "manup" about their health and prevents them from taking care of their diabetes. This study examines how we can assist Black men in improving their diabetes. Based on the traits of John Henry, we will conduct a culturally-tailored study to 1) determine if our education program including coping strategies and motivation text messages lowers A1c; and, 2) how program operates in a rural setting while learning how we can best improve it for a larger study. We hope to have the information to conduct a larger study with Black men in rural areas to improve their diabetes outcomes.

DETAILED DESCRIPTION:
As the United States' 7th leading cause of death, improving diabetic outcomes is a public health priority. Black American men disproportionately suffer from diabetes more than White counterparts. John Henryism endorses traditional masculine norms for Black Men, such as self-determination and strength, as assets. However, these norms can also act as barriers to diabetes self-management as they restrict access to support from family and friends at a time when it is most needed.

The purpose of this application is to pilot a targeted, culturally-tailored, diabetes self-management intervention for 50 rural Black men to improve diabetes-related outcomes. Aim 1: Implement a 6-month diabetes self-management intervention, grounded in John Henryism, with two arms consisting of the active intervention group and a delayed intervention group to test the intervention's effect on the primary outcome of A1c change. Aim 2: Determine the feasibility of conducting a 6-month culturally-tailored diabetes self-management intervention for Black men in a rural NC community.

The intervention includes a 10-week education program focusing on self-management, social support and coping strategies; and, daily motivational text messages. Aim 1 analysis includes repeated measures t-test (or the non-parametric equivalent Wilcoxon Matched Pairs test) to compare the mean scores of the both groups pre and post intervention. Aim 2 analysis focuses on key parameters required for conducting a future trial. This innovative study leverages the self-reliance and active coping mechanisms of John Henryism by fostering self-determination to properly self-manage diabetes while providing stress management and coping skills to buffer John Henryism's adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1) reside in Halifax, County or Alamance County NC; 2) age 21 or older; (3) English language proficient; 4) able to walk unaided; 4) self-reported type 2 diabetes diagnosis.

Exclusion Criteria:

* Exclusion criteria includes being non-ambulatory or having a diagnosis that would preclude them from participating in an exercise program.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 1) reside in Halifax or Alamance Counties in NC; 2) age 21 or older; (3) English language proficient; 4) able to walk unaided; 4) self-reported type 2 diabetes diagnosis.
Enrollment: 50 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
A1c | 6 months
  Hemoglobin A1c (determine diabetes status over previous 2 months)

CONTACTS AND LOCATIONS:
Locations (1):
- North Carolina Central University, Durham, North Carolina, United States